CLINICAL TRIAL: NCT06886347
Title: Penpulimab Plus Gemcitabine and Anlotinib in the Treatment of Metastatic Nasopharyngeal Cancer, A Single Arm, Open-label, Phase Ib Clinical Trial
Brief Title: Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chen Xiaozhong (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaozhong, chief physicians, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-Ib-02
Record Dates: First submitted 2023-07-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Experimental: The dosage of penplimab injection is 200 mg per session, administered on the first day of each cycle, Q3W
  Interventions: Drug: Penplimab Injection; Drug: Antitinib Hydrochloride Capsules; Drug: Gemcitabine

INTERVENTIONS:
Drug: Penplimab Injection — Penplimab Injection: Intravenous infusion of Penplimab 200 mg Q3W, with a 3-week treatment cycle.
  Anlotinib Hydrochloride Capsules: 10 mg, taken orally on an empty stomach before breakfast once a day (the daily medication time should be the same as much as possible), delivered in warm water, continuously used for 2 weeks and stopped for 1 week, with a treatment cycle of 3 weeks.
  Gemcitabine injection: Intravenous infusion of 1000mg/m2, administered on the 1st and 8th days of each cycle, 3 weeks per cycle for 4-6 cycles.
Drug: Antitinib Hydrochloride Capsules — 10 mg, taken orally on an empty stomach before breakfast once a day (the daily medication time should be the same as much as possible), delivered in warm water, continuously used for 2 weeks and stopped for 1 week, with a treatment cycle of 3 weeks.
Drug: Gemcitabine — Intravenous infusion of 1000mg/m2, administered on the 1st and 8th days of each cycle, 3 weeks per cycle for 4-6 cycles.

SUMMARY:
To evaluaate the efficacy and safety of the regimen incuding Penpulimab, Gemcitabine and Anlotinib in the treatment of metastatic nasopharyngeal carcinoma. Using Progression-Free-Survival as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. The participants voluntarily signed an informed consent form.
2. Age of ≥ 18 years and ≤ 75 years at the time of enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. xpected survival of ≥ 3 months.
5. Histologically or cytologically confirmed diagnosis of stage IVb NPC (AJCC 8th).
6. Metastatic NPC patients who have not recieved the first-line platinumbased chemotherapy.
7. At least one measurable tumor lesion per RECIST 1.1 criteria.
8. Adequate organ function.
9. Female participants of childbearing potential must agree to use contraception (such as intrauterine device, contraceptive pill, or condom) during the study and for 6 months after the end of the study; must have a negative serum pregnancy test within 7 days before study entry and must not be lactating. Male participants must agree to use contraception during the study and for 6 months after the end of the study.
10. The subjects are willing and able to comply with the visit schedule, treatment plan, laboratory examination, and other requirements of the study.

Exclusion Criteria:

1. ubjects have had another malignancy within 3 years before the first dose, except nasopharyngeal carcinoma. Subjects with other malignancies that have been cured by local therapy such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervix or breast carcinoma in situ are not excluded.
2. Participation in treatment with an investigational drug or use of an investigational device within 4 weeks before first study dosing.
3. Palliative local treatment was performed for non target lesions within 2 weeks before the first administration; Received nonspecific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc., excluding IL-11 for the treatment of thrombocytopenia) within 2 weeks before the first administration; Received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week before the first administration.
4. Progression during or within 6 months after receiving systemic treatment for locally advanced disease (including induction therapy, concurrent radiotherapy, adjuvant therapy) (excluding oral single agent chemotherapy maintenance).
5. Patients with local recurrence and distant metastasis after radical treatment for locally advanced disease.
6. Patients with recurrent nasopharyngeal lesions after radiotherapy and who have received secondary radiotherapy.
7. Have previously received immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists , immune cell therapy, and other treatments against tumor immune mechanism.
8. Previously received anti angiogenic therapy.
9. According to the judgment of the investigator, there are subjects with concomitant diseases that seriously endanger the safety of subjects or affect the completion of the study, or subjects who believe that there are other reasons that are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Baseline up to 2 years
  PFS defined as the time from the first dose until the first documented progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | Baseline up to 2 years
  Percentage of subjects achieving complete response (CR) and partial response (PR)
Disease Control Rate (DCR) | Baseline up to 2 years
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD)
Overall survival (OS) | Baseline up to 2 years
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up
Time to Response (TTR) | Baseline up to 2 years
  TTR defined as the time from randomization to the first recorded CR or PR
Duration of Response (DOR) | Baseline up to 2 years
  DOR defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first.
PD-L1 expression | Tumor tissue samples must be provided to the research center prior to initial administration
  Evaluating the correlation between PD-L1 expression and efficacy in tumor tissue samples.
Blood EBV level | Baseline up to 2 years
  Evaluate the correlation between the copy number of EBV DNA in the blood of subjects and their efficacy.
Evaluate the health-related quality of life (HRQoL) of subjects | Baseline up to 2 years
  Evaluate the health-related quality of life (HRQoL) of subjects using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire scale。The minimum values is 1，the maximum values is 4，and whether higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China